CLINICAL TRIAL: NCT00063050
Title: Healthy Children Healthy Families
Brief Title: Osteoporosis Prevention: Changes to Exercise and Diet in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Melbourne Hovell, Director of CBEACH, Distinguished Professor of Public Health, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD037749 (NIH)
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Osteoporosis
Keywords: Bone density; Children; Adolescents; Behavior; Health education; Health promotion; Physical fitness; Diet; Parent training; Injury control
MeSH Terms: conditions — Osteoporosis; Behavior; Health Education | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Physical activity and nutrition intervention

SUMMARY:
The purpose of this study is to determine whether educating parents about health and behavior management techniques will increase physical activity, calcium intake, fitness, and bone density in their children.

DETAILED DESCRIPTION:
In recent years, osteoporosis has become a major public health problem in the United States. Osteoporosis can best be prevented by optimizing bone mineral gain and reducing bone loss. Because the rate of bone development reaches its peak during adolescence, fostering bone health in childhood is of critical importance. Although there have been many studies of exercise and nutritional factors that influence bone mass in adults, few randomized, prospective studies have been conducted in children. This study will determine whether parent training is effective in increasing children's calcium intake, strength, and frequency of aerobic exercise.

Families will be randomly assigned to either the physical activity and nutrition intervention group or to the injury prevention control group. Families in both groups will undergo training during 9 weekly classes. The intervention training will emphasize health topics, principles of behavior, and contingency management techniques. Post-training coaching procedures will be provided periodically for 9 months. Coaching procedures will assist parents with problem solving and help them refine and maintain parenting skills. All families will be assessed prior to training and at Months 3, 9, and 12. Outcome measures will include 24-hour recall estimates of change in diet and change in physical activity. Total bone calcium, bone density, body composition, and skeletal age will also be assessed.

ELIGIBILITY:
Inclusion Criteria

* Participates in organized sports less than 3 days a week and less than 9 months per year
* Parent willing to attend weekly training sessions

Exclusion Criteria

* Serious medical illness
* Spends less than 4 days a week with the parent willing to attend classes
* Body mass index > 32

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2000-04; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
DXA - at baseline and 9 months
Nutrient Intake Interview - at baseline, 3, 9 and 12 months
Physical Activity Recall - at baseline, 3, 9 and 12 months
Strength/Fitness measures - at baseline, 3, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Melbourne F. Hovell, Ph.D., MPH, Principal Investigator — San Diego State University
Locations (1):
- The Center for Behavioral Epidemiology and Community Health at the Graduate School of Public Health at San Diego State University, San Diego, California, United States

REFERENCES:
- [Background] Schmitz KE, Hovell MF, Nichols JF, Irvin VL, Keating K, Simon GM, Gehrman C, Jones KL. Validation study of adolescents' puberty self-assessments. Journal of Early Adolescence 2004; 24(4): 357-384.
- [Background] Nichols JF, Irvin V, Schmitz KE, Hovell MF. Body Composition and Fat Distribution in Non-Hispanic White and Hispanic Pre-Adolescents. Int J of Body Comp Res 6(1):9-16, 2008.
- [Result] Hovell MF, Nichols JF, Irvin VL, Schmitz KE, Rock CL, Hofstetter CR, Keating K, Stark LJ. Parent/Child training to increase preteens' calcium, physical activity, and bone density: a controlled trial. Am J Health Promot. 2009 Nov-Dec;24(2):118-28. doi: 10.4278/ajhp.08021111. PMID 19928484